CLINICAL TRIAL: NCT05456841
Title: Empathic Communication Skills Training to Reduce Lung Cancer Stigma
Brief Title: Empathic Communication Skills (ECS) Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); Go2 Foundation for Lung Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-339
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: lung cancer; thoracic oncology physician; thoracic oncology nurse practitioner; thoracic oncology physicians assistant; 21-339; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oncology Care Providers/OCP-intervention group (Experimental): Providers participate in Empathic Communication Skills (ECS) training
  Interventions: Behavioral: Empathic Communication Skills (ECS) training
- Oncology Care Providers/OCP-control group (Active Comparator): Providers complete all study measures and are offered ECS training after data collection is completed at their site.
  Interventions: Other: Standard of Care participant interaction
- Participants with Lung Cancer-intervention group (Experimental): Participants will engage with oncology care providers/OCP who have undergone Empathic Communication Skills (ECS) training
  Interventions: Behavioral: Empathic Communication Skills (ECS) training
- Participants with Lung Cancer-control group (Active Comparator): Waitlist control group - WLC
  Interventions: Other: Standard of Care participant interaction

INTERVENTIONS:
Behavioral: Empathic Communication Skills (ECS) training — The overall training goal of this 2.25 hour module ECS module is to enhance OCP recognition and responsiveness to lung cancer patients' empathic opportunities by communicating understanding, alleviating stigma and distress, and providing support. The ECS training also provides tools to OCPs to buffer/inoculate patients against stigmatizing attitudes and behaviors by others such that lung cancer patients who currently or formerly smoked can be given "small doses" of an opposing viewpoint (termed as "preparing patients for recurring smoking questions") and suggestions of "counterarguments" in order to make them resistant to future stigmatizing attacks by others
  Arms: Oncology Care Providers/OCP-intervention group; Participants with Lung Cancer-intervention group
Other: Standard of Care participant interaction — Standard of Care participant interaction
  Arms: Oncology Care Providers/OCP-control group; Participants with Lung Cancer-control group

SUMMARY:
Research indicates that perceived stigma within medical encounters is prevalent and problematic for lung cancer patients' well-being and quality of cancer care. Promoting empathic communication appears to be a potentially effective intervention target to help reduce patients' perceptions of stigma within clinical encounters; however, no formal trainings exist that focus on teaching empathic communication to oncology care providers (OCPs). Building upon favorable findings from a prior R21 (R21CA202793) and the importance of developing interventions to address lung cancer stigma, our goal is to conduct a national trial of empathic communication skills (ECS) training to facilitate improvements in the medical and psychosocial care of patients through de-stigmatizing interactions with OCPs for patients diagnosed with lung cancer.

DETAILED DESCRIPTION:
The aims of this study are:

1. to evaluate the effect of the ECS training on OCP primary outcomes (communication and empathic skill uptake) and secondary outcomes (ECS training appraisal - relevance, novelty, clarity; self-efficacy, empathy, compassion burn-out);
2. to evaluate the effect of the ECS training vs. WLC on patients' reported primary outcomes (lung cancer stigma), and secondary outcomes (perceived clinician empathy, satisfaction with communication, psychological distress, patients' experience of clinical encounter, and overall patient satisfaction).

   Additionally, acceptance of referral to tobacco cessation (for those currently smoking) will be explored; and
3. to examine potential moderators of OCP (e.g., demographic characteristics, professional role characteristics) and patient outcomes (e.g., demographic characteristics, illness characteristics).

Our central hypothesis is that the ECS training will demonstrate significant short-term improvements in clinicians' uptake of empathic skills and self-efficacy and will be superior to WLC with regards to patient reported measures of stigma, clinician empathy, satisfaction, and overall experience.

ELIGIBILITY:
Inclusion Criteria:

Site Eligibility

* Employs at least 15 FTE OCPs (i.e., oncologists, nurse practitioners and physician assistants) as per self report
* Reports a clinic volume of at least 20 new lung cancer patients per month as per self report

OCP Participant Eligibility

* OCPs who are thoracic oncology physicians (radiologists, medical oncologists, pulmonologists, and surgeons), NPs, or PAs and currently treating lung cancer patients, as per self-report;
* OCP conducts consultations with lung cancer patients, as per self-report;
* OCP sees at least 1 lung cancer patient per week, as per self-report;

Patient Eligibility

* Patient under the care of a participating OCP as per self report;
* English and/or Spanish speaking;

  * In general, which language do you prefer to receive your medical care, English/Spanish/both English and Spanish Equally?
  * If English, treat as fluent in English, no additional language questions
  * If Spanish, treat as fluent in Spanish, no additional language questions
  * If both English and Spanish equally, ask the follow-up questions and go with whichever language is endorsed as best. If endorsed equally, assign to category patient prefers
  * How well do you speak English? Not at all/ Not well/Well/Very well
  * How well do you speak Spanish? Not at all/Not well/Well/Very well
* Is at least 18 years of age as per self report;
* Has a history of suspicious lung mass or confirmed lung cancer diagnosis, as per clinician judgment or medical record note;
* Is a former or current smoking as per self report;
* Has had no more than 10 prior visits with the participating OCP, as per the medical record and/or self report

Exclusion Criteria:

Patient Exclusion

* Individuals of impaired decision-making capacity as per a clinician's judgment or as documented in the EMR.

Site and OCP Exclusion

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1232 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of communication skills using standardized patient assessment/SPAs | 3 months
  A SPA involves a 12-minute video recorded interaction between the Oncology Care Provider/OCP and the Standardized Patient/SP on a given clinical scenario, using standardized scripts by the SP. Each OCP will participate in one SPA prior to their ECS training and one SPA following training or the timed control period. In contrast to clinical consultation recordings with varied clinical situations that do not necessitate the use of all strategies and skills, the semi-structured nature of SPAs permits appraisal of all desired elements of training.
Uptake of empathy skills using standardized patient assessment/SPAs | 3 months
  A SPA involves a 12-minute video recorded interaction between the Oncology Care Provider/OCP and the Standardized Patient/SP on a given clinical scenario, using standardized scripts by the SP. Each OCP will participate in one SPA prior to their ECS training and one SPA following training or the timed control period. In contrast to clinical consultation recordings with varied clinical situations that do not necessitate the use of all strategies and skills, the semi-structured nature of SPAs permits appraisal of all desired elements of training.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Banerjee, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Providence St. Joseph Health (Data Collection Only), Irvine, California
  - BAPTIST ALLIANCE - MCI (Data Collection Only), Miami, Florida
  - Advocate Health Care Network, Libertyville, Illinois
  - University of Kentucky (Data Collection Only), Lexington, Kentucky
  - Munson Healthcare (Data Collection Only), Traverse City, Michigan
  - Hackensack Meridian Health (Data collection only), Hackensack, New Jersey
  - Roswell Park Cancer Institute (Data Collection Only), Buffalo, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Virtua Health (Data Collection Only), Philadelphia, Pennsylvania
  - University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania
  - Chesapeake Regional Healthcare (Data Collection Only), Chesapeake, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Banerjee SC, Malling CD, Schofield EA, Carter-Bawa L, Bylund CL, Hamann HA, Parker PA, Shen MJ, Studts JL, Williamson TJ, Ostroff JS. Empathic communication skills training to reduce lung cancer stigma: Study protocol of a cluster randomized control trial. Contemp Clin Trials. 2024 Oct;145:107669. doi: 10.1016/j.cct.2024.107669. Epub 2024 Aug 23. PMID 39182827
- [Derived] Banerjee SC, Malling CD, Shen MJ, Williamson TJ, Bylund CL, Studts JL, Mullett T, Carter-Bawa L, Hamann HA, Parker PA, Steliga M, Feldman J, Pantelas J, Borondy-Kitts A, Rigney M, King JC, Fathi JT, Rosenthal LS, Smith RA, Ostroff JS. Getting ready for prime time: Recommended adaptations of an Empathic Communication Skills training intervention to reduce lung cancer stigma for a national multi-center trial. Transl Behav Med. 2023 Sep 28;13(10):804-808. doi: 10.1093/tbm/ibad048. PMID 37579304
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org